CLINICAL TRIAL: NCT04168710
Title: Ultrasound Guided Emergency Physician Performed Erector Spinae Nerve Block for Rib Fracture Analgesia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000025328; No NIH funding (Other: 12.19.23)
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The clinical team taking care of the patient as well as the patient will be blinded as to allocation to experimental or control group. The physician administering the block will also be blinded to the substance administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- erector spinae plane block (ESP block) with bupivacaine (Experimental): Each participant randomized to the ESP block group will receive an ultrasound guided single shot injection of 20cc of 0.25% bupivacaine in the plane between the transverse process of the spine and the erector spinae muscle.
  Interventions: Drug: ESP block with bupivacaine
- ESP block with saline/sham injection (Placebo Comparator): Each participant randomized to the ESP block group will receive an ultrasound guided single shot injection of 20cc of normal saline in the plane between the transverse process of the spine and the erector spinae muscle.
  Interventions: Other: Saline control/sham injection

INTERVENTIONS:
Drug: ESP block with bupivacaine — Each participant randomized to the ESP block group will receive an ultrasound guided single shot injection of 20cc of 0.25% bupivacaine in the plane between the transverse process of the spine and the erector spinae muscle.
  Arms: erector spinae plane block (ESP block) with bupivacaine
Other: Saline control/sham injection — Each participant randomized to the ESP block group will receive an ultrasound guided single shot injection of 20cc of normal saline in the plane between the transverse process of the spine and the erector spinae muscle.
  Arms: ESP block with saline/sham injection

SUMMARY:
The study will be a prospective randomized double blinded placebo controlled clinical trial using ultrasound guided erector spinae plane block as an analgesic adjunct among adult emergency department (ED) patients with rib fractures using mean morphine milligram equivalents as the primary outcome.

DETAILED DESCRIPTION:
Aim 1: Given the novelty of the erector spinae plane nerve block and limited data from anesthesia literature, aim 1 is to obtain preliminary data regarding quantity of mean morphine equivalents received by control and experimental groups for an initial subset of 50 patients to improve sample size calculation and better power the study.

Aim 2: Evaluate efficacy of ED performed ultrasound guided ESP block in delivering analgesia by evaluating difference in morphine milligram equivalents (MME) as well as pain scores during ED stay and hospital admission between the experimental and control groups.

Aim 3: Evaluate adverse event rates related to ultrasound guided ESP block placement as well as rates of rib-fracture related complications between control and experimental groups.

ELIGIBILITY:
Inclusion Criteria:

1. radiographic evidence of unilateral rib fracture(s).
2. able to consent and actively participate in the study.
3. moderate to severe pain (defined as numerical pain rating score >/ 4 ) at time of enrollment.

Exclusion Criteria:

1. known allergy or hypersensitivity to local anesthetics or morphine.
2. infection at site of ESP block placement.
3. depth over 5 cm from skin to transverse process visualized with ultrasound.
4. additional injuries that preclude positioning for ESP block placement.
5. severe traumatic brain or spinal cord injury.
6. severe altered mental status, such that pain could not be assessed.
7. extra thoracic injuries for which rib pain is reported as less than the rest of the injuries.
8. adjunctive epidural catheter pain control.
9. other regional anesthetic blocks.
10. pregnancy or prisoner status.
11. unstable vital signs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Total intravenous (IV) and oral narcotic analgesic use | From enrollment/baseline in the study through the study period, up to 24 hours.
  narcotic use will be measured in morphine milligram equivalents (MME), based on dosing and frequency.

SECONDARY OUTCOMES:
Pain score | Baseline (immediately following recruitment).
  Pain scores will be measured using a standard11-point numerical rating scale that ranges from 0 ("no pain") to 10 ("worst pain imaginable)
Pain score | 30 minutes post-baseline
  Pain scores will be measured using a standard11-point numerical rating scale that ranges from 0 ("no pain") to 10 ("worst pain imaginable)
Pain score | 1 hour post-baseline
  Pain scores will be measured using a standard11-point numerical rating scale that ranges from 0 ("no pain") to 10 ("worst pain imaginable)
Pain score | 4 hours post-baseline
  Pain scores will be measured using a standard11-point numerical rating scale that ranges from 0 ("no pain") to 10 ("worst pain imaginable)
Pain score | 12 hours post-baseline
  Pain scores will be measured using a standard11-point numerical rating scale that ranges from 0 ("no pain") to 10 ("worst pain imaginable)
Pain score | 24 hours post-baseline
  Pain scores will be measured using a standard11-point numerical rating scale that ranges from 0 ("no pain") to 10 ("worst pain imaginable)
Hospital length of stay (LOS) | From hospital admission to hospital discharge, up to 30 days.
  LOS will be identified through the electronic medical record.
Number of Patients Who Develop Pneumonia | From admission to 30 days from admission.
  Identified through review of the electronic medical record for a discharge diagnosis of pneumonia, or readmission diagnosis of pneumonia within 1 month from presentation.
Adverse events associated with the nerve block itself. | Within two hours of administration of the nerve block.
  Adverse events will include: hypotension, respiratory depression, and nausea or vomiting. Hypotension will be defined as a systolic blood pressure < 90 mmHg and respiratory depression as respiratory rate < 10 breaths per minute. Nausea or vomiting will be defined as patient-reported sensation of nausea or actual emesis, documented emesis in the medical record, or administration of an antiemetic during the study period.
Total non-narcotic analgesic use. | From enrollment/baseline in the study through the study period, up to 24 hours.
  Non-narcotic analgesic use will be measured by medical record review of all non-narcotic medications. Groups will be compared with respect to each category: non-steroidal anti-inflammatory use, acetaminophen use, local anesthetic patch use.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiana Baloescu, MD, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No